CLINICAL TRIAL: NCT03024398
Title: Evaluation of the Fluorescent Green of Indocyanine in the Detection of Sentinel Lymph Node in Endometrial Cancer
Acronym: Sentimetre
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6492
Record Dates: First submitted 2017-01-05; First posted 2017-01-18 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cancer of the Endometrium
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Selective lymphadenectomy Sentinel (LSS). This technique is already well established in breast cancer and melanoma and more recently in vulvar and cervical cancer.

Compared to lymphadenectomy, it has several theoretical advantages:

* this is a sensitive technique with a detection rate of> 90% and a false negative rate of <5%.
* the anatomopathological techniques used (immunohistochemistry with anti-cytokeratin antibodies, serial sections) are more sensitive than the standard histological analysis of lymphadenectomy, which allows an improvement in the detection of metastases (micro-metastases, isolated tumor cells). In the SENTI-ENDO study, it was possible to detect lymph node metastases in 11% of patients with low-risk endometrial cancer and in 15% of intermediate-risk patients.
* it avoids short-term and long-term operative and post-operative morbidity of lymphadenectomy.

Early studies of LSS in endometrial cancer demonstrated superior efficacy of the colorimetric method coupled with the Technetium 99m isotopic method with an overall detection rate of 78% [95% CI: 73-84]. The fluorescent green of indocyanine appears to give better results with an overall detection rate of 94% and a bilateral detection rate of 80%.

It seemed useful to take stock of this technique using this new dye.

ELIGIBILITY:
Inclusion Criteria:

* Major patient, without guardianship or curatorship.
* patient with endometrial cancer confirmed by biopsy.
* Invasive cancer stage FIGO I at intermediate risk and high risk and II according to the FIGO classification.
* need for surgical staging.
* performing an endovaginal ultrasound or a pelvic MRI in preoperative, if contraindication to MRI, performing a CT scan.
* subject affiliated to a social health insurance scheme.
* speaking and reading French.
* subject having dated and signed informed consent.

Exclusion Criteria:

* pregnancy in progress.
* FIGO III and IV stage diagnosed preoperatively or intraoperatively.
* Cure or pre-surgery that may alter the uterine lymphatic drainage (conization, myomectomy).
* MRI or CT scan of suspected lymph nodes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with confirmed biopsy endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Detection of sentinel node | 1 hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cherif Youssef AKLADIOS, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de gynécologie-obstétrique - Hôpital de Hautepierre, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No